CLINICAL TRIAL: NCT06791824
Title: A Phase IB/II Clinical Study to Assess the Safety, Tolerability and Preliminary Efficacy of CM313(SC) Injection in Subjects With Relapsed/Refractory Aplastic Anemia
Brief Title: Study of CM313(SC) Injection in Subjects With Relapsed/Refractory Aplastic Anemia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CM313-124101
Record Dates: First submitted 2025-01-15; First posted 2025-01-24 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CM313(SC)(low dose group) (Experimental)
  Interventions: Biological: CM313(SC) injection
- CM313(SC)(medium dose group) (Experimental)
  Interventions: Biological: CM313(SC) injection
- CM313(SC)(high dose group) (Experimental)
  Interventions: Biological: CM313(SC) injection

INTERVENTIONS:
Biological: CM313(SC) injection — Phase IB: CM313(SC) administered at low dose according to the protocol. Phase II: CM313(SC) administered at different doses based on Phase IB's results.
  Arms: CM313(SC)(low dose group)
Biological: CM313(SC) injection — Phase IB: CM313(SC) administered at medium dose according to the protocol. Phase II: CM313(SC) administered at different doses based on Phase IB's results.
  Arms: CM313(SC)(medium dose group)
Biological: CM313(SC) injection — Phase IB: CM313(SC) administered at high dose according to the protocol. Phase II: CM313(SC) administered at different doses based on Phase IB's results.
  Arms: CM313(SC)(high dose group)

SUMMARY:
This is a randomized, open-label, phase IB/II clinical study to evaluate the safety, tolerability and preliminary efficacy of CM313(SC) injection in patients with relapsed/refractory aplastic anemia

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of idiopathic aplastic anemia.
2. Patients must meet the requirements of relapsed/refractory aplastic anemia defined in the protocol.
3. Male or female, age≥18 years.
4. The Eastern Cooperative Oncology Group (ECOG) physical status score ≤2.
5. Willing and able to comply with the requirements for this study and written informed consent.

Exclusion Criteria:

1. The inherited bone marrow failure syndromes.
2. Previously treated with the anti-CD38 monoclonal antibody.
3. Have an allergy to humanized monoclonal antibody or any part of CM313.
4. Pregnant or breastfeeding females, or females planning to become pregnant during the study.
5. Any condition considered to be ineligible for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Estimated)
Dates: Start 2025-03 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AE) | Up to 52 weeks
  Assess the safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Jun Shi, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China